CLINICAL TRIAL: NCT00444145
Title: Do Laryngeal Biopsy Findings Predict Treatment Response in Suspected Laryngopharyngeal Reflux
Brief Title: Do Laryngeal Tissue Changes in Patients Suspected of Having Laryngopharyngeal Reflux Predict Response to Treatment?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 061244
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Larynx Disease; Gastroesophageal Reflux
MeSH Terms: conditions — Laryngeal Diseases; Gastroesophageal Reflux | interventions — Lansoprazole; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with documented GERD or laryngopharyngeal reflux (Experimental): Patients who have documented GERD as evidenced by erosive esophagitis or those patients who have newly diagnosed laryngopharyngeal reflux as diagnosed by endoscopy.
  Interventions: Drug: Prevacid; Procedure: Esophageal and Laryngeal Biopsies

INTERVENTIONS:
Drug: Prevacid — 30 mg bid for 3 months
  Other Names: lansoprazole
Procedure: Esophageal and Laryngeal Biopsies — repeat egd with biopsy after Prevacid 30 mg bid for 3 months
  Other Names: esophagogastroduodenoscopy

SUMMARY:
The purpose of the study is to determine if tissue changes are predictor of clinical response to therapy.

The hypothesis is that the patients who have laryngeal signs and symptoms related to acid reflux, will have ultrastructural changes on a laryngeal biopsy which are predictors of response to therapy.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) has been implicated, in part, as the cause of various laryngeal signs and symptoms (1-7). This is often termed reflux laryngitis, ear, nose, and throat (ENT) reflux, or laryngopharyngeal reflux (LPR). GERD was first described to be a causative agent in developing contact ulcers of the larynx (8), and since this early report other routinely observed laryngeal signs are now attributed to LPR. These include laryngeal edema/erythema, vocal cord granulomas and polyps, posterior cricoid cobblestoning, interarytenoid changes, and subglottic stenosis. In addition, patient symptoms attributed to LPR include hoarseness, sore or burning throat, chronic cough, throat clearing, globus, nocturnal laryngospasm, otalgia, post-nasal drip, and dysphagia.

GERD occurs in 7% - 25% of the population on a daily or monthly basis, respectively (9). It is estimated that up to 10% of patients presenting to ENT physicians do so because of complaints that are thought to be related to LPR (2).

The current management of patients with suspected LPR complaints include either 1. empiric therapy using proton pump inhibitors (PPI's) or 2. Ambulatory 24-hour pH monitoring to test for GERD before beginning treatment. Because of the uncertainty and subjectivity of the ENT laryngeal examination in diagnosing LPR, both algorithms fall short of ideal in treating these patients. In a recent review of the literature, remarkably, up to 50% of patients with laryngoscopic signs suggesting LPR do not respond to aggressive acid suppression and do not have abnormal esophageal acid reflux values on pH testing (10). Yet, in this subset of patients LPR continues to be implicated as the probable etiology of the patient's laryngeal signs and symptoms.

Calabrese, et al. recently looked at the reversibility of GERD related ultrastructural alterations in the esophagus using a PPI. Lower esophageal biopsies were analyzed with electron microscopy (EM) for ultrastructural alterations attributed to GERD; that is, dilation of intracellular spaces. Patients were then treated with a PPI and re-biopsied for analysis of any changes of healing that may have occurred in these ultrastructural alterations. Not surprisingly, the ultrastructural alterations showed complete recovery (reduction of dilated intracellular spaces) after treatment with a PPI. Additionally resolution of patient's symptoms coincided with recovery of ultrastructural alterations (11). No such biopsies looking for LPR related changes in the larynx have ever been performed in human subjects. Our initial study which is also submitted for review will provide data on the prevalence of biopsy findings in controls, GERD and LPR patients. Subsequent to this prevalence study, the importance of these findings will be assessed based to determine if these findings will predict response to acid suppressive therapy.

In sum, LPR is an extremely subjective diagnosis, in which nearly half of all patients do not have an abnormal 24hr pH study, nor do they respond to the standard GERD therapy of acid suppression. Finding an alternative objective criterion for GERD induced laryngitis would be an important clinical discovery. To date, there are no data on microscopic changes in the larynx of patients suspected of having LPR. The most important question which this protocol will address is if laryngeal findings specifically by either routine microscopy or electron microscopy would predict response to PPI therapy. This would then result in being able to identify GERD related laryngitis from non-GERD related causes.

ELIGIBILITY:
Inclusion Criteria:

GERD

* Documented erosive esophagitis:

  * Patients will be newly diagnosed with esophageal erosion at initial visit via EGD
  * Patients with non-erosive esophagitis who have been responsive to PPI

LPR

* Diagnosed via Head & Neck Institute endoscopists:

  * pts with chronic (> 3-months) history of hoarseness, throat clearing, sore- or burning throat and globus
  * Documentation of LPR using Larynx/Pharynx exam.

This group is commonly evaluated at the Vanderbilt Voice Center.

Exclusion Criteria:

* Age < 18yrs
* Pregnancy
* Patients with contra-indications for EGD
* Patients on corticosteroids
* Active smokers
* Patients with a history of regular (> 2 /day) alcohol use.
* Use of antacid (PPI, H2RB) within last 30 days
* Use of any/all medications affecting gastrointestinal motility
* Known history of: Barrett's esophagus, Peptic stricture, Pyloric stenosis, Gastric resection
* Patients unable to give informed consent
* Patients unable to comply with follow-up
* Patients with known contraindication to lansoprazole.
* Contraindications to biopsy: Taking anticoagulants other than aspirin (Coumadin, Plavix) or allergic to the local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD,PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Endoscopy Lab, TVC 1410, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Prevacid: Patients who have documented GERD as evidenced by erosive esophagitis or those patients who have newly diagnosed laryngopharyngeal reflux as diagnosed by endoscopy.
  Prevacid: 30 mg bid for 3 months
  Esophageal and Laryngeal Biopsies: repeat egd with biopsy
Period: Overall Study
Arm/Group | Patients Receiving Prevacid
Started | 38
Completed | 19
Not Completed | 19
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — non-compliant | 11
Not completed — Screen Failures | 5

BASELINE CHARACTERISTICS:
Population: Patients diagnosed with GERD as evidenced by erosive esophagitis and patients diagnosed with laryngopharyngeal reflux (LPR)
Arm/Group | Patients Receiving Prevacid
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dilation of Intracellular Spaces 3 Months After Therapy
Description: Dilation of inter cellular spaces (the space within the cell) is reported to be an early morphological (structure and form) marker in gastro-oesophageal reflux. Using electron microscopy, the distance between epithelial cells is quantified.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Patients Receiving Prevacid
Number analyzed (Participants) | 19
participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Patients Receiving Prevacid
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes